CLINICAL TRIAL: NCT06066294
Title: A Randomized Controlled Trial on Safety and Immunogenicity of Purified Verocell Rabies Vaccine as Pre-exposure Prophylaxis Via Intradermal Two Visits (2-0-2-0-0) Verses Three Visits (1-0-1-0-1) Regimen on Healthy Volunteers
Brief Title: A Comparison of Safety and Immunogenicity of Rabies Pre Exposure Prophylaxis Regimen Between Gvt of India Approved and WHO Approved.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kempegowda Institute of Medical Sciences, Bangalore (Other Government)
Responsible Party: Principal Investigator, Dr. N.R. Ramesh Masthi, Professor and Head of Department, Department of Community Medicine, Kempegowda Institute of Medical Sciences, Bangalore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KIMSCM01
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Vaccine Reaction
Keywords: Immunogenicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regimen 1 (Experimental): WHO recommended PrEP Vaccination Schedule, 2 visits, 0.2ml 2 sites (0.1ml each site) on day 0 and day 7
  Interventions: Biological: Regimen 1
- Regimen 2 (Active Comparator): Government of India currently recommended PrEP Schedule, 0.1ml 3 visits, on day 0, day 7 and day 28
  Interventions: Biological: Regimen 2

INTERVENTIONS:
Biological: Regimen 1 — WHO Pre-qualified rabies vaccine (Rabivax-S), WHO recommended PrEP Vaccination Schedule, 2 visits, 0.2ml 2 sites (0.1ml each site) on day 0 and day 7
  Arms: Regimen 1
Biological: Regimen 2 — WHO Pre-qualified rabies vaccine (Rabivax-S), Government of India approved vaccination schedule, 3 visits, 0.1ml 1 site on day 0, 7 and 28
  Arms: Regimen 2

SUMMARY:
The goal of this clinical trial is to compare WHO recommended PrEP Vaccination Schedule, 2 doses 0.2ml 2 sites (0.1ml each site) on day 0 and day 7 and Government of India currently recommended PrEP Schedule, 0.1ml 3 doses on day 0, day 7 and day 28 in Healthy subjects above 18years of age, willing to volunteer and sign written informed consent for the study. The main questions it aims to answer are:

* To assess the seroconversion (? 0.5 IU/mL) of the study subjects following primary & boosting vaccination on Day 35 ,Day 365, Day 372/375.
* To assess the incidence of adverse events(immediate/delayed, local/systemic) among subjects.

Participants will be administerd with WHO Pre-qualified rabies vaccine (Rabivax-S) .

Researchers will compare the two regimens mentioned above.

DETAILED DESCRIPTION:
The study will be conducted among healthy adult volunteers visiting the Anti Rabies Clinic, Preventive Medicine Unit, Kempegowda Institute of Medical Sciences Hospital& Research Centre, Bangalore and visits to other institutes/places in bangalore.

Step-1: Selection of Volunteers: The healthy volunteers who agreed to participate in the study will be screened for the inclusion and exclusion criteria and subsequently explained regarding the vaccination regimen, benefits due to vaccine and informed consent will be taken. The selected volunteers will be randomized into two groups-study and control group.

Step-2: Collection of Data: A pre tested semi structured questionnaire will be used for collection of data about Socio demographic profile and other related variables.

Step-3: Vaccination of Volunteers: The volunteers will be given WHO Pre-qualified rabies vaccine (Rabivax-S, purchased from open market) 0.1ml each in 2 sites on Day 0 & 7 intradermal for the study group and 0.1 ml of rabies vaccine at 1 site intradermal route on Day 0, 7 & 28 for the control group. Later, in each group, 50% of the subjects will be provided a booster dose of vaccine i.e. 0.1 ml, one site on day 365(one visit); for another 50 % of the subjects, booster dose of vaccine i.e. 0.1 ml, one site on days 365 and 368(two visits).

Step 4: Safety evaluation: After each vaccination dose, subject will be observed for an hour, to find out any adverse drug reactions (ADRs) and then, a follow-up card will be given to enter any ADRs during the entire period of vaccination and one week after the last dose. All the reported ADRs will be recorded and analysed. The adverse events will be classified according to the revised adverse events following immunization (AEFI) guidelines.12 Step 5: Collection of Sample and immunogenicity analysis: 5ml of venous blood will be collected from the ante-cubital vein on day-0 (before vaccination), day-35 (after last dose of vaccination) and day 365. For subjects who have received 0.1 ml booster dose on day 365, 5ml blood sample will be collected on day 372 and for those subjects, who have received 0.1ml booster dose on day 365 and 368, 5ml blood sample will be collected on day 375 to estimate rabies virus neutralizing antibody(RVNA) titres. The samples collected from the volunteers are centrifuged, serum separated and stored in -200 Centigrade at the Anti Rabies Clinic, Preventive Medicine Unit, Kempegowda Institute of Medical Sciences Hospital& Research Centre, Bangalore. The serum will be transported in cold chain to the Department of Neurovirology, National Institute of Mental Health and Neuro Sciences, Bangalore which is the WHO collaborating centre for reference and research on rabies, where the Rapid fluorescent focus inhibition test (RFFIT) is done to estimate RVNA titres. The results obtained from RFFIT will be shared to the volunteers. Information regarding next dose and sample collection will be given to the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects willing to volunteer and sign written informed consent for the study.
* Subjects should be available for the follow-up period.

Exclusion Criteria:

* Received Anti rabies vaccine or RIG or RMAb anytime in the past.
* Participation in any other clinical trial in the past three months.
* Severely immunocompromised subjects, pregnant and lactating women.
* Subjects with known history of allergy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
To assess the seroconversion (>0.5 IU/mL) of the study subjects following primary & boosting vaccination on Day 35 ,Day 365, Day 372/375. | Blood samples will be collected on Day 0, Day 35, Day 365, Day 372 and Day 375
  5ml of venous blood will be collected from the ante-cubital vein on day-0 (before vaccination), day-35 and day 365. For subjects who have received 0.1 ml booster dose on day 365, 5ml blood sample will be collected on day 372 and for those subjects, who have received 0.1ml booster dose on day 365 and 368, 5ml blood sample will be collected on day 375 to estimate rabies virus neutralizing antibody(RVNA) titres. The Rapid fluorescent focus inhibition test (RFFIT) is done at the Department of Neurovirology, National Institute of Mental Health and Neuro Sciences, Bangalore which is the WHO collaborating centre for reference and research on rabies, to estimate RVNA titres. The results obtained from RFFIT will be shared to the volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Deekshith J Reddy, MBBS, Principal Investigator — Kempegowda Institute of Medical Sciences
Locations (1):
- Kempegowda Institute Of Medical Sciences Hospital and Research Center, Bengaluru, Karnataka, India